CLINICAL TRIAL: NCT04014777
Title: A Phase 1, Multicenter, Open-Label, Single-Dose and Multiple-Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Intravitreal Injections of NGM621 in Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: Study of NGM621 in Participants With Geographic Atrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-0501
Record Dates: First submitted 2019-07-03; First posted 2019-07-10 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NGM621 Cohort 1 Single Ascending Dose (Experimental): NGM621 single IVT injection Cohort-Dose 1
  Interventions: Biological: NGM621
- NGM621 Cohort 2 Single Ascending Dose (Experimental): NGM621 single IVT injection Cohort--Dose 2
  Interventions: Biological: NGM621
- NGM621 Cohort 3 Single Ascending Dose (Experimental): NGM621 single IVT injection Cohort--Dose 3
  Interventions: Biological: NGM621
- NGM621 Cohort 4 Multiple Dose (Experimental): NGM621 multiple IVT injection Cohort--Dose 4
  Interventions: Biological: NGM621

INTERVENTIONS:
Biological: NGM621 — NGM621 Dose 1
  Arms: NGM621 Cohort 1 Single Ascending Dose
Biological: NGM621 — NGM621 Dose 2
  Arms: NGM621 Cohort 2 Single Ascending Dose
Biological: NGM621 — NGM621 Dose 3
  Arms: NGM621 Cohort 3 Single Ascending Dose
Biological: NGM621 — NGM621 Dose 4
  Arms: NGM621 Cohort 4 Multiple Dose

SUMMARY:
This is a multi-center evaluation of NGM621 in an open-label, single-dose and multiple-dose escalation study in participants with Geographic Atrophy secondary to Age-related Macular Degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. GA lesion size in the study eye of >=2.5 mm² as assessed by the central reading center
2. BCVA - 54 to 4 letters (20/80 to 20/400 Snellen equivalent) using the standard ETDRS (Early Treatment of Diabetic Retinopathy Study) in the study eye at the Screening and Baseline visits; the fellow eye must have a BCVA of at least 69 letters (Snellen equivalent 20/40) at the Screening and Baseline visits

Exclusion Criteria:

1. GA in either eye because of cause other than AMD
2. History or evidence of glaucoma or ocular hypertension in either eye as defined by investigator
3. Visual impairment in the study eye due to causes other than GA
4. Spherical equivalent of the refractive error in the study eye demonstrating more than -6 Diopters of myopia (prior to cataract or refractive surgery)

Other protocol-defined inclusion/exclusion criteria could apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Ocular and Systemic Treatment-Emergent Adverse Events (TEAEs) | 12 weeks
  The number and percent of patients reporting treatment emergent adverse events (TEAEs) by cohort.

SECONDARY OUTCOMES:
Serum Concentration of NGM621 | 12 weeks
  Individual and mean serum NGM621 concentration data by cohort.

CONTACTS AND LOCATIONS:
Overall Officials: NGM Study Director, Study Director — NGM Biopharmaceuticals
Locations (6):
- United States (6):
  - NGM Clinical Study Site, Arcadia, California
  - NGM Clinical Study Site, Newport Beach, California
  - NGM Clinical Study Site, Melbourne, Florida
  - NGM Clinical Study Site, St. Petersburg, Florida
  - NGM Clinical Study Site, Austin, Texas
  - NGM Clinical Study Site, The Woodlands, Texas